CLINICAL TRIAL: NCT06851897
Title: Comparison of Perforated 3D Printed Metal Fixed Mandibular Retainer Versus Conventional Fixed Bonded Retainer A Randomized Clinical Trial
Brief Title: Comparison of Perforated 3D Printed Versus Conventional Metal Fixed Bonded Retainer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mariam Alaa (Other)
Responsible Party: Sponsor-Investigator, Mariam Alaa, Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Orth 332; Cairo University (Other: Cairo University)
Record Dates: First submitted 2025-02-12; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Bond, Pair
MeSH Terms: conditions — Pair Bond

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional fixed retainer (Active Comparator): multistrand or braided metal wire
  Interventions: Other: conventional fixed retainer
- Perforated 3D printed metal fixed retainer (Experimental): 3D printed wire custom made to each patient after intraoral scanning
  Interventions: Other: perforated 3D printed metal fixed retainer

INTERVENTIONS:
Other: perforated 3D printed metal fixed retainer — The key of modification is digitally designing fixed metal retainer which will be custom made for each patient, and 3D metal printing of the fixed retention wire using Metal printer instead of using generic metal wire for all patients.
  Arms: Perforated 3D printed metal fixed retainer
Other: conventional fixed retainer — Conventional fixed metal retainer will be used. Multi strand wire will be used
  Arms: Conventional fixed retainer

SUMMARY:
Although different materials of mandibular fixed retainer were discussed in the literature, there is contradicting evidence regarding the bond failure of Titanium fixed metal retainer, whether immediate or after 12 months. Moreover, insufficient evidence is present regarding 3D metal printed fixed mandibular retainers.

DETAILED DESCRIPTION:
In recent years a new possibility is available for dental practitioners: CAD-CAM technology and 3D printing, which find their application in all aspects of orthodontics. Orthodontists are already familiar with several products that use 3D printers (i.e. invisible aligners), also known as additive manufacturing, 3D printing is a technology whereby sequential layers of material are layered on top of one another to form an object23. Two recent articles reported the fabrication of a custom lingual retainer cut from a nickel-titanium block with CAD/CAM technology and a CAD/CAM Zirconium bar as a bonded mandibular fixed retainer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with properly finished orthodontic treatment.
* No sex predilection.
* The presence of 4 permanent mandibular incisors and 2 permanent mandibular canines.
* No active caries, restorations, fractures, or periodontal disease of previously mentioned teeth
* Patients with good oral hygiene.

Exclusion Criteria:

* Patients with no need of fixed mandibular retention.
* Enamel hypoplasia or hypocalcification of mandibular anterior teeth.
* Abnormal morphology of mandibular anterior teeth
* Periodontal disease that contraindicates fixed orthodontic retention.
* No or poor patient's compliance & bad oral hygiene.
* Psychological problems.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Bond Failure | immediate up to 12 months
  Counting number of teeth debonded immediately after placement of wire up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariam MA Elsebaey, Phd, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT06851897/Prot_SAP_ICF_000.pdf